CLINICAL TRIAL: NCT02406872
Title: A Study Comparing Remimazolam Tosilate and Propofol for Intravenous General Anaesthesia in Operations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HR7056-002
Record Dates: First submitted 2015-02-15; First posted 2015-04-02 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Remimazolam Tosilate 1 (Experimental): IV pumping of Remimazolam Tosilate at 6mg/kg/h for anesthesia induction
  Interventions: Drug: Remimazolam Tosilate
- Remimazolam Tosilate 2 (Experimental): intravenous pumping of Remimazolam Tosilate at 12mg/kg/h for anesthesia induction
  Interventions: Drug: Remimazolam Tosilate
- Remimazolam Tosilate 3 (Experimental): intravenous pumping of Remimazolam Tosilate at 18mg/kg/h for anesthesia induction
  Interventions: Drug: Remimazolam Tosilate
- Propofol (Active Comparator): single IV bolus of Propofol at 2.0-2.5mg/kg for anesthesia induction
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Tosilate — IV pumping for anesthesia
  Arms: Remimazolam Tosilate 1; Remimazolam Tosilate 2; Remimazolam Tosilate 3
Drug: Propofol — IV bolus for anesthesia
  Arms: Propofol

SUMMARY:
The purpose of this study is to find out the optimal dose for Remimazolam Tosilate as an intravenous general anaesthetic drug in operations and to determine its efficacy and safety profile comparing to propofol.

DETAILED DESCRIPTION:
This is an multi-center，double-blinded，parallel and control study using Remimazolam or propofol for anesthesia in operations.Subjects are randomized to different treatment groups (including 3 for Remimazolam Tosilate and 1 for propofol) and anaesthetics are pumped contimuously into bodies.Analgesics and muscle relaxants are permitted during operations.Efficacy，safety and pharmacokinetic/pharmacodynamic profiles of Remimazolam Tosilate are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18-60 years；
* intending to have non-emergency operations；
* ASA( American Society of Anesthesiologists) I or II；
* 18 kg/m²<BMI(Body Mass Index)<30 kg/m².

Exclusion Criteria:

* people with contraindications to general anaesthesia;
* one or more of the laboratory findings fall out of the limitations for this study(platelet,hemoglobin,aspartate aminotransferase,etc.);
* history of recent use of narcotics,analgesics,anaesthetics and benzodiazepine hypnotics;
* history of severe cardiovascular disease;
* uncontrolled blood glucose level;
* cerebral disease or mental disorder;
* allergic to drugs used in the study;
* pregnant women or those in lactation period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
successful anaesthesia rate as measured by the proportion of subjects who experienced succesful anesthesia during operations | an average of 3 hours (immediately after opaerations)

SECONDARY OUTCOMES:
bispectral index(BIS) during anaesthesia as measured by bispectral index machine | every 5 minutes
recovery time as measured by time | an average of 3 hours (after cessation of anesthetics pumping)
induction time as measured by time | 1-10 minutes (from the begining of anesthetics)

OTHER OUTCOMES:
rate of improper-depths sedation as measured by the proportion of subjects who experienced too-deep or too-shallow anesthesia during operations | an average of 3 hours (after anesthesia)
rate of hypotention as measured by the proportion of subjects who experienced hypotention during operations | an average of 3 hours (after anesthesia)
rate of hyoxemia as measured by the proportion of subjects who experienced hyoxemia during operations | an average of 3 hours (after anesthesia)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China